CLINICAL TRIAL: NCT00875875
Title: Single Daily Dose Rifaximin vs. Standard Thrice Daily Dosing for the 3-Day Treatment of Travelers' Diarrhea
Brief Title: Single Daily Dose Rifaximin for the Treatment of Travelers' Diarrhea
Acronym: Rifaximin 600
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No study population in Mexico (H1N1). Study withdrawn from IRB consideration.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Charles D Ericsson, ◦Professor and Dr. and Mrs. Carl V. Vartian Professor in Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ericsson-001
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Travelers' Diarrhea
Keywords: Diarrhea, travelers; Acute travelers' diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): This is the approved treatment regimen for travelers' diarrhea (600 mg)
  Interventions: Drug: Rifaximin
- 2 (Active Comparator): This is the same dose as the standard dose, given once daily (200 mg)
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 200 mg TID for 3 days OR Rifaximin 600 mg Daily for 3 days
  Other Names: Xifaxin

SUMMARY:
The study will compare durations of diarrhea among subjects who report to clinic for treatment and who receive either:

1. standard rifaximin therapy at a dose of 200 mg three times a day for 3 days, OR
2. a single 600 mg dose of rifaximin daily for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* passage of 3 or more unformed stools in 24 hours plus an additional symptom of enteric disease such as abdominal cramps, nausea, vomiting, or fever; and investigator verification that an unformed stool has been submitted.
* is > 18 years of age
* has diarrhea (at least three unformed stools in 24 hrs) plus at least one additional sign or symptom of enteric illness
* has acute diarrhea less than 1 week's duration
* willingness to provide a diarrhea stool sample
* willingness to keep a daily diary for 5 days
* signed informed consent

Exclusion Criteria:

* fever or bloody diarrhea
* has taken predictably effective antibiotics in the past week (e.g. quinolones, TMP/SMX, azalide or doxycycline)
* is pregnant now, likely to become pregnant, or breast-feeding
* has duration of diarrhea of greater than 1 weeks
* is allergic to Rifampin or Rifaximin
* has a history of significant underlying enteric, pulmonary, cardiac, renal disease, or any CNS disorder
* is more than moderately dehydrated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Time from beginning therapy to passage of last unformed stool | 5 days

SECONDARY OUTCOMES:
Side effects as reported by the subjects on diaries | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Ericsson, MD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- Enteric Disease Clinic, Guadalajara, Jalisco, Mexico